CLINICAL TRIAL: NCT01326520
Title: Effect of Dietary Milk Phospholipids on Subjects With Atopic Dermatitis
Brief Title: Effect of Dietary Phospholipids on Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LSEP H49-11
Record Dates: First submitted 2011-03-28; First posted 2011-03-31 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phospholipid enriched dairy product (Experimental)
  Interventions: Dietary Supplement: milk phospholipid
- dairy product (Placebo Comparator)
  Interventions: Dietary Supplement: diary product

INTERVENTIONS:
Dietary Supplement: milk phospholipid — The patients will consume daily 250 mL of a dairy product, which is enriched with 3 g of milk phospholipids.
  Arms: Phospholipid enriched dairy product
Dietary Supplement: diary product — The patients will consume daily 250 mL of a common dairy product.
  Arms: dairy product

SUMMARY:
The aim of the study is to investigate the influence of a milk phospholipid enriched dairy product on subjects with atopic dermatitis determining parameters of the immune status, the plasma lipid profile and the skin texture.

DETAILED DESCRIPTION:
Based on the facts, that on the one hand milk phospholipids are characterized by a high sphingolipid content and on the other hand a disturbed sphingolipid metabolism in the epidermis of patients with atopic dermatitis was verified, a double blinded, controlled, randomized, cross-over study with a daily supplementation of 3 g milk phospholipids to subjects with a mild to moderate atopic dermatitis will be conducted.

Forty patients will be randomized between two groups of each 20 patients. After an individual checkup and a run-in period of 2 weeks, the one group will receive the phospholipid enriched dairy product and the second group will be given a placebo dairy product over two month. A wash out-period of 4 weeks will follow, and the patients will consume the contrary dairy products over two month after a 2-week run-in period again.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate atopic dermatitis (SCORAD < 30)
* age: 18 - 60 years

Exclusion Criteria:

* intolerance against milk proteins
* systemic medication with corticosteroids or antihistamines
* immune mediated disease
* atherosclerosis
* hyperlipidaemia
* diabetes mellitus
* angina pectoris
* adipositas
* pregnancy and breast feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in skin texture from baseline and in comparison with placebo | after 0,2,10,16, and 24 weeks
  SCORAD Index

SECONDARY OUTCOMES:
Immune status | after 0,2,10,16, and 24 weeks
  total IgE, specific IgE, sE selectin, Interferon-gamma, Tumor necrosis factor-alpha, Interleukin 4, 12, 16, 31
Lipid status | after 0,2,10,16, and 24 weeks
  Blood lipids (Total cholesterol, LDL cholesterol, HDL cholesterol, triacyl glycerdies, fatty acids, phospholipids)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller Univesity of Jena, Department of Nutritional Physiology
Locations (1):
- Friedrich Schiller University Jena, Department of Nutritonional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Keller S, Le HY, Rodiger C, Hipler UC, Kertscher R, Malarski A, Hunstock LM, Kiehntopf M, Kaatz M, Norgauer J, Jahreis G. Supplementation of a dairy drink enriched with milk phospholipids in patients with atopic dermatitis - a double-blind, placebo-controlled, randomized, cross-over study. Clin Nutr. 2014 Dec;33(6):1010-6. doi: 10.1016/j.clnu.2014.01.014. Epub 2014 Jan 29. PMID 24559855